CLINICAL TRIAL: NCT00113438
Title: A Randomized Open-Labeled Phase II Study of Combretastatin A-4 Phosphate in Combination With Paclitaxel and Carboplatin to Evaluate the Safety and Efficacy in Subjects With Advanced Imageable Malignancies
Brief Title: Safety and Effectiveness of Combretastatin A-4 Phosphate Combined With Chemotherapy in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA4P-212; HCI-13214 (Other: Huntsman Cancer Institute)
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Cancer; Tumor
Keywords: cancer; tumor; imageable; CA4P; Combretastatin; Combretastatin A4 Phosphate; Combretastatin A-4 Phosphate; Carboplatin; Paclitaxel; carbo; taxol
MeSH Terms: conditions — Neoplasms | interventions — fosbretabulin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 45 mg/m2 Combretastatin A-4 Phosphate (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate + Paclitaxel + Carboplatin
- 60 mg/m2 Combretastatin A-4 Phosphate (Experimental)
  Interventions: Drug: Combretastatin A-4 Phosphate + Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Combretastatin A-4 Phosphate + Paclitaxel + Carboplatin — Combretastatin A-4 Phosphate is administered IV at 45 mg/m2 or 60 mg/m2 on Days 1, 8 and 15 followed by paclitaxel (3 hour infusion at 200 mg/m2) and carboplatin (1 hour infusion at AUC = 6) on Day 2 of each cycle. The treatment cycle is 21 days with a maximum of 21 days. Following cycle 6, subjects that have not progressed may continue on CA4P monotherapy, which will be administered at 45 mg/m2 or 60 mg/m2 on Days 1 and 8 with rest on Day 15, repeated every 21 days until disease progression.
  Other Names: CA4P; fosbretabulin; paclitaxel; carboplatin

SUMMARY:
This is a study evaluating the safety and effectiveness of Combretastatin A4 Phosphate (CA4P) combined with the chemotherapy drugs, carboplatin and paclitaxel. The full treatment and observation time should be about 5 months. During this time the patient should receive 18 CA4P infusions and 6 carboplatin followed by paclitaxel treatments. Patients will be randomized into one of two CA4P dose-level groups in order to recommend a preferred dose-level for future studies. At least 2 dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) scans will be conducted to monitor the blood flow through the tumor before and after treatment with CA4P.

DETAILED DESCRIPTION:
This is a phase II study evaluating the safety and efficacy of Combretastatin A4 Phosphate (CA4P) combined with carboplatin and paclitaxel. Treatment is for a maximum of 6 consecutive 21-day cycles. Patients are randomized onto one of two CA4P dosing arms (45 or 63 mg/m2). CA4P is administered on days 1, 8 and 15 of each cycle. Carboplatin and paclitaxel (AUC 6 and 200 mg/m2, respectively) are administered on day 2 of each cycle. At least 2 DCE-MRI scans will be performed to evaluate the change in tumor blood flow following treatment with CA4P.

ELIGIBILITY:
Inclusion Criteria:

* Advanced malignancy where treatment with carboplatin and paclitaxel is warranted.
* Minimum 28-day interval from any surgical, chemotherapy or immunotherapy treatment and a 14-day interval from radiotherapy treatment.
* Radiologically measurable disease to meet MRI perfusion criteria.
* ECOG performance status less than or equal to 1.
* Life expectancy greater than 12 weeks.
* Normal ejection fraction.

Exclusion Criteria:

* Uncontrolled brain metastasis.
* Significant cardiac abnormalities.
* Prior radiotherapy at the tumor site.
* Symptomatic peripheral vascular or cerebrovascular disease.
* Uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To assess safety of the CA4P-paclitaxel-carboplatin combination in advanced imageable malignancies | From first administration of study drug through approximately 30 days following last dose of study drug
To evaluate tumor response | From baseline through end of study visit
To establish the Recommended Phase II Dose (RP3D) for the combination of CA4P-paclitaxel-carboplatin in advanced imageable malignancies | from first study drug administration through end of study visit
To assess the change in tumor blood flow by use of MRI in advanced imageable malignancies | from screening through end of study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States